CLINICAL TRIAL: NCT02443285
Title: Is Spontaneous Bacterial Peritonitis Still Responding to 3rd Generation Cephalosporins?
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sherief Abd-Elsalam, PI, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SBP TREATMENT
Record Dates: First submitted 2015-05-11; First posted 2015-05-13 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Primary Bacterial Peritonitis
MeSH Terms: interventions — Cefotaxime; Ceftriaxone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cefotaxime (Active Comparator): cefotaxime 2gm every 12 hours daily for 5 days
  Interventions: Drug: Cefotaxime
- Ceftriaxone (Active Comparator): ceftriaxone 2 gm every 24 hours for 5 days.
  Interventions: Drug: ceftriaxone

INTERVENTIONS:
Drug: Cefotaxime — Cefotaxime 2 gram every12 hours for 5 days
  Other Names: claforan, cefotax
  Arms: Cefotaxime
Drug: ceftriaxone — Ceftriaxone 2 gm every 24 hours for 5 days
  Other Names: rocephin, cefaxone
  Arms: Ceftriaxone

SUMMARY:
Current European and most other international guidelines recommend the use of a third-generation cephalosporin as the first choice, or amoxicillin-clavulanate acid or fluoroquinolones as an alternative choice .

These recommendations are based mainly on clinical trials that were very often conducted a decade or more ago, and on the assumption that E. coli would be involved in nearly half of the cases.

The microbial etiology of SBP remains relatively constant; however, the antibiotic resistance rate especially for third-generation cephalosporins (including cefotaxime and ceftazidime), ciprofloxacin, and ofloxacin increased dramatically .

DETAILED DESCRIPTION:
Spontaneous bacterial peritonitis (SBP), defined as an infection of ascites in the absence of a contiguous source of infection.

Spontaneous bacterial peritonitis (SBP) is a common and potentially fatal bacterial infection in patients with cirrhosis and ascites, occurring in 10 to 30% of patients, with in-hospital mortality rates ranging from 20 to 30% .

It is secondary to impaired humoral and cellular immune responses that result in indirect intestinal bacterial translocation into the ascitic fluid .

SBP is also associated with a poor long-term prognosis for patients, as mortality rates can reach 50 to 70% at 1 year .

Early diagnosis and early optimal treatment of these infections with appropriate antibiotics and the prevention of hepatorenal syndrome with albumin are required .

Current European and most other international guidelines recommend the use of a third-generation cephalosporin as the first choice, or amoxicillin-clavulanate acid or fluoroquinolones as an alternative choice.

These recommendations are based mainly on clinical trials that were very often conducted a decade or more ago, and on the assumption that E. coli would be involved in nearly half of the cases.

The microbial etiology of SBP remains relatively constant; however, the antibiotic resistance rate especially for third-generation cephalosporins (including cefotaxime and ceftazidime), ciprofloxacin, and ofloxacin increased dramatically.

ELIGIBILITY:
Inclusion Criteria:

* Liver cirrhosis with ascites and SBP

Exclusion Criteria:

* ascitic fluid with polymicrobial infections

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
number of patients with clearence of infection | 5 days
  number of patients having clearence of infection

CONTACTS AND LOCATIONS:
Overall Officials: Sherief M Abd-elsalam, lecturer, Principal Investigator — hepatology dept-Tanta; Hanan H Soliman, Professor, Study Director — hepatology dept-Tanta; Walaa A Elkhalawany, lecturer, Study Chair — hepatology dept-Tanta
Locations (1):
- Tanta university - faculty of medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided